CLINICAL TRIAL: NCT01308788
Title: Examination of the Effect of Aqueous Suppressant Versus Aqueous Outflow Enhancing Glaucoma Medications on Ocular Perfusion Pressure and Blood Flow: A Mechanistic Study
Brief Title: Aqueous Suppressant Versus Aqueous Outflow on Ocular Blood Flow
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: IGPS-prost-OAG
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Glaucoma
Keywords: glaucoma blood flow
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- aqueous suppressant: aqueous suppressant treated
- aqueous outflow: aqueous outflow treated

SUMMARY:
The purpose of this study will be to compare the aqueous production suppressant to aqueous outflow drugs in terms of the response to known vascular parameters. Specifically; systemic perfusion pressure, retrobulbar blood flow and retinal microcirculation.

DETAILED DESCRIPTION:
The purpose of this study will be to compare the aqueous production suppressant to aqueous outflow drugs in terms of the response to known vascular parameters. Specifically; systemic perfusion pressure, retrobulbar blood flow and retinal microcirculation.

A comparison of perfusion pressure, retinal microcirculation utilizing Heidelberg Retinal Flowmetry and retrobulbar circulation utilizing color Doppler ultrasound imaging

ELIGIBILITY:
Inclusion Criteria:

Patients will meet all of the following inclusion criteria to enter the study:

1. Age: 30 years or older.
2. Diagnosis: confirmed open-angle glaucoma in at least one eye:

   1. glaucomatous visual field loss on Humphrey 24-2 or 10-2 perimetry
   2. glaucomatous optic disc cupping
   3. agreement between two baseline exams for reliability
3. Best corrected visual acuity at least 20/60 in at least one eye.
4. Prior Humphrey visual fields demonstrate acceptable reliability standards (see below).

Exclusion Criteria:

1. Extensive Humphrey visual field damage consisting of either a mean deviation (MD) < -15 decibels or a clinically determined threat to fixation in both hemifields.
2. Evidence of exfoliation or pigment dispersion.
3. History of acute angle-closure or a narrow, occludable anterior chamber angle by gonioscopy.
4. History of chronic or recurrent inflammatory eye diseases (e.g., scleritis, uveitis).
5. History or signs of intraocular trauma.
6. Severe or potentially progressive retinal disease such as retinal degeneration, diabetic retinopathy, and retinal detachment.
7. Any abnormality preventing reliable applanation tonometry.
8. Current use of any ophthalmic or systemic steroid which may interfere with this investigation.
9. Cataract surgery within the past year.
10. Resting pulse < 50 beats per minute.
11. Severe, unstable or uncontrolled cardiovascular, renal, or pulmonary disease.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 glacuoma patients
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alon Harris, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Department of Ophthalmology Indiana University School of Medicine, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recited over 6 months
Period: 6-month Treatment
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Started | 14 | 21
Completed | 14 | 21
Not Completed | 0 | 0
Period: 2-year Treatment
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Started | 14 | 21
Completed | 10 | 10
Not Completed | 4 | 11
Not completed — medication change by treating physician | 4 | 11

BASELINE CHARACTERISTICS:
Population: There will be (as shown) differences in the number of subjects based upon the time of analysis due to patient loss, data of insufficient quality at visit, or change in the drug use during period of study (patient switched off treatment by their doctor) so the number of data points varies throughout the analysis by availability.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aqueous Suppressant | Aqueous Outflow | Total
Number analyzed (Participants) | 21 | 14 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 12 | 6 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 21 | 14 | 35

OUTCOME MEASURES:

1. Primary Outcome: 6-month Change in Ophthalmic Artery (OA) Peak Systolic Velocity (PSV)
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 14 | 21
cm/sec | -.70 (2.57) | 1.84 (.96)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .4414, ANCOVA

2. Primary Outcome: 6-month Change in Phthalmic Artery (OA) End Diastolic Velocity (EDV)
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 14 | 21
cm/sec | -.36 (.78) | .12 (.44)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .7820, ANCOVA

3. Primary Outcome: 6-month Change in Phthalmic Artery (OA) Vascular Resistance (RI)
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 14 | 21
unitless | .003 (.011) | .014 (.013)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .5496, ANCOVA

4. Primary Outcome: 6-month Change in Central Retinal Artery (CRA) Peak Systolic Velocity (PSV)
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 14 | 21
cm/sec | -.16 (.28) | .09 (.25)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .2930, ANCOVA

5. Primary Outcome: 6-month Change in Central Retinal Artery (CRA) End Diastolic Velocity (EDV)
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 14 | 21
cm/sec | -.13 (.10) | -.03 (.11)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .5058, ANCOVA

6. Primary Outcome: 6-month Change in Central Retinal Artery (CRA) Vascular Resistance (RI)
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 14 | 21
unitless | .029 (.018) | .005 (.010)
Statistical Analysis 1: Comparison: Aqueous Outflow; Test type: Superiority or Other; p = .6156, ANCOVA

7. Primary Outcome: 6-month Change in Ocular Perfusion Pressures (OPP)
Time Frame: Baseline and 6 month visits
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 14 | 21
mm Hg | -3.38 (2.26) | -.63 (2.36)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .5443, ANCOVA

8. Primary Outcome: 2-year Change in OA PSV
Time Frame: Baseline and 24 month visits
Population: one participant was unable to be measured for this outcome
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 10 | 9
cm/sec | 1.39 (3.05) | 2.63 (3.40)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .7847, ANCOVA

9. Primary Outcome: 2-year Change in OA EDV
Time Frame: Baseline and 24 month visits
Population: one participant was unable to be measured for this outcome
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 10 | 9
cm/sec | -1.28 (.71) | .34 (.62)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .1331, ANCOVA

10. Primary Outcome: 2-year Change in OA RI
Time Frame: Baseline and 24 month visits
Population: one participant was unable to be measured for this outcome
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 10 | 9
unitless | .035 (.016) | .019 (.029)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .5431, ANCOVA

11. Primary Outcome: 2-year Change in CRA PSV
Time Frame: Baseline and 24 month visits
Population: one participant was unable to be measured for this outcome
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 10 | 9
cm/sec | 1.46 (.64) | .19 (.50)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .0684, ANCOVA

12. Primary Outcome: 2-year Change in CRA EDV
Time Frame: Baseline and 24 month visits
Population: one participant was unable to be measured for this outcome
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 10 | 9
cm/sec | .43 (.24) | .16 (.33)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .2500, ANCOVA

13. Primary Outcome: 2-year Change in CRA RI
Time Frame: Baseline and 24 month visits
Population: one participant was unable to be measured for this outcome
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 10 | 9
unitless | .005 (.017) | -.010 (.030)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .6896, ANCOVA

14. Primary Outcome: 2-year Change in OPP
Time Frame: Baseline and 24 month visits
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Number analyzed (Participants) | 10 | 10
mm Hg | -1.26 (3.36) | -3.02 (4.69)
Statistical Analysis 1: Comparison: Aqueous Outflow vs Aqueous Suppressant; Test type: Superiority or Other; p = .7965, ANCOVA

ADVERSE EVENTS:
Description: Adverse events were not assessed/collected as a part of this study protocol
Arm/Group | Aqueous Outflow | Aqueous Suppressant
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Small number of subjects at final endpoint, participation number various by analysis and date

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No